CLINICAL TRIAL: NCT04175938
Title: Assessment of Corneal Endothelial Function Following Hypoxic Stress
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Ula Jurkunas, Associate Professor, Harvard Medical School, Massachusetts Eye and Ear Infirmary
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019P002073
Record Dates: First submitted 2019-11-18; First posted 2019-11-25 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Fuchs' Endothelial Corneal Dystrophy
Keywords: Fuch's Dystrophy, FECD, Fuch's Endothelial Corneal Dystrophy
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Intervention Model Description: A stress test will be performed (the wearing of a contact lens) to induce swelling in two groups: group A where the subjects have a diagnosis of Fuch's Endothelial Corneal Dystrophy, and group B where subjects have healthy eyes. Once the contact lens is removed, the cornea swelling will be measured in each group. The length of time it takes for the cornea to recover after being swollen will also be compared between the two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Subjects with Fuch's Endothelial Dystrophy (Active Comparator): Persons with a diagnosis of Fuch's Endothelial Dystrophy will wear a contact lens in an affected eye for three hours.
  Interventions: Device: Wearing of contact lens
- Subjects with healthy eyes (Other): Persons with healthy eyes will wear a contact lens in one eye for three hours.
  Interventions: Device: Wearing of contact lens

INTERVENTIONS:
Device: Wearing of contact lens — All subjects will wear a contact lens for three hours. The effect of the lens on the eye (epithelial swelling) will be measured at intervals after the lens is removed.

SUMMARY:
The purpose of this study is to determine the difference in the cornea's response to contact lens placement between healthy and unhealthy eyes. The amount of corneal swelling (corneal thickness) between normal and FECD patients before and after a stress test will be measured and compared.

DETAILED DESCRIPTION:
Clarity of the cornea is essential for optimal vision. The endothelium is a layer within the cornea that controls its clarity. Fuchs endothelial corneal dystrophy (FECD) is a progressive disease that affects both eyes in which the endothelium is dysfunctional, causing the cornea to swell and lose its clarity. Because of the vision loss associated with this swelling, corneal transplantation is needed for patients with advanced FECD.

Currently, there is no method to directly measure how well endothelium cells are functioning in patients with FECD. Such a measurement, if it were possible, would allow physicians to identify patients who are at a higher risk of corneal swelling. The goal of this study is to establish a tool to measure and compare the amounts of corneal swelling between normal and FECD patients after a stress test is performed (the wearing of an FDA-approved contact lens.) Data will also be collected regarding how quickly and how well a cornea recovers from swelling in patients with healthy eyes compared to those with FECD.

ELIGIBILITY:
Inclusion Criteria:

Subjects in the Fuch's Dystrophy arm of the study must meet following criteria:

* Have a clinical diagnosis of Fuchs endothelial corneal dystrophy
* Be scheduled for corneal transplantation in the next 6 months
* Have no history of prior ocular surgery in study eye
* Have no history of contact lens intolerance
* Be motivated and willing to complete ocular imaging tests

Subjects in the healthy eyes arm of the study must meet following criteria:

* Have no prior history of ocular disease including ocular surface disease or glaucoma
* Have no history of prior ocular surgery in study eye
* Have no history of contact lens intolerance
* Be motivated and willing to complete ocular imaging tests

Exclusion Criteria: Pregnant women

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Thickness of the cornea before and after the stress test | seven hours
  Maximum changes in the thickness of the cornea measured before and after the stress test
The rate of corneal recovery after the stress test | three hours
  The extent of swelling evident at regular intervals during the 3 hours after the stress test
Time to full recovery from swelling | three hours
  The time it takes for the eye to no longer be swollen

CONTACTS AND LOCATIONS:
Overall Officials: Ula Jurkunas, MD, Principal Investigator — Massachusetts Eye and Ear
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States